CLINICAL TRIAL: NCT04381533
Title: Internet-based Adolescent Community Reinforcement Approach (I-A-CRA) With Therapist Support for Young Adults With Problematic Alcohol Use: A Randomized Controlled Trial
Brief Title: Internet-based A-CRA for Young Adults With Problematic Alcohol Use
Acronym: I-A-CRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nitya Jayaram-Lindstrom (Other)
Responsible Party: Sponsor-Investigator, Nitya Jayaram-Lindstrom, Principal Investigator, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1264-31/5
Record Dates: First submitted 2020-04-28; First posted 2020-05-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Abuse; Binge Drinking; Alcohol Use Disorder
Keywords: Randomized Controlled Trial; Alcohol; Internet-delivered Psychological Treatment; Behavior Therapy; Young Adults
MeSH Terms: conditions — Alcoholism; Binge Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-A-CRA (Experimental): Internet-delivered Adolescent Community Reinforcement Approach: The treatment program consists of 8 extensive treatment modules delivered over 10 weeks with continuous therapist support and guidance. There are two separate treatments for the young adult and the caregiver/significant other.
  Interventions: Behavioral: Internet-delivered Adolescent Community Reinforcement Approach (I-A-CRA)
- Psychoeducation alcohol use (Active Comparator): Psychoeducation focusing on alcohol use: This support program provides 8 brief modules of psychoeducation (alcohol information) over 10 weeks. Participants receive no therapist guidance/support but have the possibility of asking questions to a therapist. There are two separate programs for the young adult and the caregiver/significant other.
  Interventions: Behavioral: Psychoeducation, information on use of alcohol and its effects

INTERVENTIONS:
Behavioral: Internet-delivered Adolescent Community Reinforcement Approach (I-A-CRA) — The intervention is a behavioral internet-based intervention based on the Adolescent Community Reinforcement Approach. The program encompasses text, pictures, videos, and written as well as practical assignments (skills training). The main components of the treatment for the young adult with problematic alcohol use consist of psychoeducation and functional analysis, goal formulation, increasing prosocial behaviors, relapse prevention, problem solving, and communication training. The accompanying significant other receives modules containing information focusing on gaining an understanding of the treatment components aimed at the young adult, as well as communication training to improve communication between the young adult and the significant other.
  Arms: I-A-CRA
Behavioral: Psychoeducation, information on use of alcohol and its effects — The intervention is a behavioural internet-based intervention including psychoeducation focusing on providing information on alcohol, alcohol use, and its effects. The psychoeducation is provided via texts and pictures, and there is a possibility of asking questions to a therapist if needed however no therapist contact is mandatory. There are separate programs directed towards the young adult and the accompanying significant other. The programmes give brief self-help tips at the end. The intervention approximately corresponds to the information given in a primary care setting for someone with problematic alcohol use.
  Arms: Psychoeducation alcohol use

SUMMARY:
The primary aim of the study is to evaluate the feasibility and acceptability of an internet-delivered Adolescent Community Reinforcement Approach (I-A-CRA) with therapist support for young adults (aged 18-24 years) with problematic alcohol use and their caregiver/significant other. Secondary aims include investigating the role of comorbid emotional symptoms, emotion regulation and prosocial behavior in treatment outcomes for the young adults. In a randomized controlled pilot trial, participants (n = 60 young adults as well as an optional accompanying caregiver/significant other) will be recruited from the community through advertisements as well as through clinic referrals in Stockholm, Sweden. Eligible participants will be randomized either to the 10-week I-A-CRA treatment or to an active control group (receiving psychoeducation about alcohol use over the same time frame). In both conditions an optionally accompanying caregiver/significant other will receive a support program in conjunction with the young adult's treatment. Participating young adults will be evaluated with regards to their alcohol use, psychiatric symptoms, emotion regulation, and prosocial behavior at pre-treatment, weekly during treatment, post-treatment, and at a 3-month follow-up. The primary outcome will be feasibility (measured as number of treatment completers; i.e., having completed 5 out of 8 treatment modules), and acceptability (measured by patient satisfaction). Secondary outcomes will include pre- and post-treatment self-rated binge drinking episodes, levels of depression, anxiety and stress, emotion dysregulation, and prosocial behavior. Self-reports regarding stress, emotion dysregulation, and prosocial behavior will be complemented by behavioral measures (computerized tasks).

ELIGIBILITY:
Inclusion Criteria:

* Young adult between 18-24 years of age
* Reporting ongoing substance use (alcohol), heavy drinking measured as risky use according to recommendations: 5/4 (male/female) standard drinks on a minimum of two occasions in the last month, or AUDIT-C ≥ 4 points indicating harmful consumption
* Access to internet via computer or other similar device, as well as access to smartphone
* If on psychiatric medication, it should have been a stable dosage during the past 3 months prior to pre-treatment assessment
* Adequate knowledge in the Swedish language and a Swedish personal identification number

Exclusion Criteria:

* Current DSM-5 diagnosis for any other substance use disorder except nicotine dependence
* Current (including last 12 months) DSM-5 diagnosis for other major psychiatric disorder (bipolar disorder, psychosis)
* Recent initiation of psychiatric medication or psychotherapy (within the last 3 months)
* Suicidal ideation at screening
* Serious somatic diagnosis requiring medical attention, such as uncontrolled diabetes mellitus, epilepsy or heart conditions
* Traces of any psychoactive substance (e.g., central stimulant amines, THC, benzodiazepines, opiates, cocaine) in urine sample at baseline assessment
* Pregnancy

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of treatment completers defined as patients completing 5 or more of the 8 modules of treatment | Will be assessed post treatment (11 weeks after treatment initiation)
  Outcome used to assess feasibility.
Client Satisfaction Questionnaire 8 item | Will be assessed post treatment (11 weeks after treatment initiation)
  Acceptance will be measured as percentage of participants rating their satisfaction as good. Higher score indicates better outcome. Scores range from 8-32.

SECONDARY OUTCOMES:
Timeline Follow-back - change in time spent doing activities unrelated to drinking | Will be assessed before treatment initiation, at week 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 of treatment, and post treatment (11 weeks after treatment initiation)
  Number of self-reported activities registered that are not related to alcohol consumption over the past week. More episodes is a better outcome.
Alcohol Use Disorders Identification Test - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-reported screening of alcohol use disorder symptoms. Higher scores indicate worse outcome. Scores range from 0-40.
Difficulties in Emotion Regulation Scale 16 item - change over timepoints | Will be assessed before treatment initiation, at week 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 of treatment, and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring emotion dysregulation. Higher scores indicate worse outcome. Scores range from 16-80.
Depression Anxiety Stress Scale-21 - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring symptoms of depression, anxiety and stress over the past week. Higher scores indicates worse outcome. Scores range from 0-42.
Timeline Follow-back - change in self-rated alcohol consumption | Will be assessed before treatment initiation, at week 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 of treatment, and post treatment (11 weeks after treatment initiation)
  Number of heavy drinking episodes (heavy drinking defined as 4 or more drinks per drinking occasion in women and 5 or more for men) over the past week. Fewer episodes is a better outcome.

OTHER OUTCOMES:
Barratt Impulsiveness Scale - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring behavioral impulsivity. Higher scores indicates worse outcome. Scores range from 30-120.
Adult ADHD Self-Report Screener - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring ADHD symptoms. Higher score indicates worse outcome.
Obsessive Compulsive Drinking Scale - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring compulsive drinking.
Pro-social behavior - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Computerized experimental behavior tasks measuring reward-based pro-social behavior and decision making regarding generous, trustful, reciprocal and compensatory behavior.
Emotion regulation/distress tolerance (Paced Auditory Serial Addition Task) - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Computerized behavior task measuring emotion regulation/distress tolerance. A longer time spent doing the task indicates better outcome.
Drinking Motive Questionnaire Revised Short Form - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring drinking motives.
Drug Use Disorders Identification Test - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report screening of any drug use disorder symptoms. Higher score indicates worse outcome. Scores range from 0-44.
Social Interaction Anxiety Scale - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring symptoms of social anxiety.
Prosocial Tendencies Measure - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring prosocial behavior.
Oxford Utilitarianism Scale - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring prosocial behavior.
Questionnaire of Cognitive and Affective Empathy - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring prosocial behavior (empathy).
Positive Personality Traits - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring prosocial behavior (positive personality traits).
Social Value Orientation - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring prosocial behavior.
Autism Spectrum Quotient Short Form - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring symptoms of autism spectrum disorder. Higher scores indicate worse outcome.
Positive and Negative Affect Schedule - Negative affect - change pre to post treatment | Will be assessed before treatment initiation and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring negative affect in the moment on a 5-point scale (higher score indicates more negative affect).
VAS Single Item Craving Question - change over timepoints | Will be assessed before treatment initiation, at week 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 of treatment, and post treatment (11 weeks after treatment initiation)
  Self-report scale measuring craving for alcohol in the moment on a visual analog scale ranging from 0-100 (a higher score indicates more craving).
Significant other, change in rating of drinking in the young adult (with Timeline Follow-back) | Will be assessed at week 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 of treatment
  Self-report scale measuring alcohol use in the young adult as assessed by significant other in the past week. Higher number of episodes indicates worse outcome.
Socioeconomic and Demographic Questionnaire | Will be assessed before treatment initiation
  Self-report of demographic information.
EQ-5D | Will be assessed before treatment initiation
  Self-report scale measuring disability (a higher score indicates worse outcome) and generic health status (rated on a visual analog scale ranging from 0-100 where higher score indicates better outcome).
Family Tree Questionnaire | Will be assessed before treatment initiation
  Self-report scale assessing family history of alcohol problems, number of family history-positive and family history-negative relatives.
Negative Effects Questionnaire | Will be assessed post treatment (11 weeks after treatment initiation)
  Self-report scale measuring negative effects associated with psychotherapy. Higher score indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nitya Jayaram-Lindstrom, Ph.D., Principal Investigator — Department of Clinical Neuroscience, Karolinska Institutet
Locations (1):
- eStod, Maria Ungdom, Stockholm Centre for Dependency Disorders, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in accordance with institutional guidelines at the Karolinska Institutet, Stockholm, Sweden.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code